CLINICAL TRIAL: NCT05957692
Title: Vitamin D and Adipose Tissue: Storage or Sequestration
Brief Title: Vitamin D and Adipose Tissue: a Complex Relationship
Acronym: ADIPOVITAD
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Principal Investigator, Luca Giuseppe Dalle Carbonare, Associate Professor, Azienda Ospedaliera Universitaria Integrata Verona
Other Study IDs: ADIPOVITAD
Record Dates: First submitted 2023-07-07; First posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Hypovitaminosis D
Keywords: vitamin D; ultrasound; adipose tissue; storage
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to verify the role of adipose tissue in determining the vitamin D serum level after monthly oral administration in subjects with vitamin D deficiency.

The main questions it aims to answer are:

* Adipose tissue represents a storage environment for vitamin D or it's an environment where vitamin D is sequestered and no longer released
* On the other hands, it's possible to verify whether the adipose tissue carries out a bi-modal activity towards vitamin D
* If adipose tissue exerts a bi-modal effect, it is possible to identify a specific threshold between the two effects Participants will undergo anthropometric measurements (height, weight, waist/hip ratio waist circumference) at baseline and after 6 months of intake of cholecalciferol 50,000 IU/month

DETAILED DESCRIPTION:
Vitamin D deficiency and insufficiency are prevalent worldwide, and various factors contribute to their occurrence, including low sun exposure, poor dietary intake, obesity, and abdominal obesity. Abdominal obesity, assessed by waist circumference (WC), is associated with metabolic syndrome and has been linked to low vitamin D levels. This study aimed to investigate the relationship between visceral adipose tissue (VAT) and vitamin D levels, particularly examining the potential threshold for vitamin D storage and sequestration by adipose tissue.

The study is conducted on patients with hypovitaminosis D in an internal medicine outpatient department. Blood samples for the evaluation of calcium and vitamin D levels are collected at baseline and after six months of monthly cholecalciferol supplementation. Ultrasonography are used to evaluate adipose tissue measurements, including subcutaneous adipose tissue thickness, VAT, preperitoneal adipose tissue (PPAT), and prerenal adipose tissue (PRAT). Anthropometric measures such as waist-to-hip ratio and waist-to-height ratio are also assessed.

ELIGIBILITY:
Inclusion Criteria:

* Vitamin D level < 20 ng/ml
* BMI > 24

Exclusion Criteria:

* Administration of vitamin D metabolites in the last year
* Previous diagnosis of metabolic bone diseases
* Previous diagnosis of endocrine diseases
* Previous diagnosis of cancer

Ages: 60 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients referred to the internal medicine clinic for cardiovascular evaluation.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline of vitamin D levels at 6 months | 6 months
  blood sample expressed in ng/ml
Change from Baseline of height measurements at 6 months | 6 months
  height expressed in cm
Change from Baseline of weight at 6 months | 6 months
  weight expressed in Kg
Change from Baseline of waist and hip circumference at 6 months | 6 months
  waist and hip circumference expressed in centimeters
Change from Baseline of body adipose tissue at 6 months | 6 months
  body adipose index expressed in percentage
Change from Baseline of ultrasound adipose tissue measurement at 6 months | 6 months
  visceral, subcutaneous, pre-renal, pre-peritoneal adipose tissue expressed in millimeters

SECONDARY OUTCOMES:
Change from Baseline of calcium levels at 6 months | 6 months
  blood sample expressed in mg/dl

CONTACTS AND LOCATIONS:
Overall Officials: Maria Teresa Valenti, BSc, Study Chair — Universita di Verona
Locations (1):
- Azienda Ospedaliera Universitaria Integrata, Verona, Italy

REFERENCES:
- [Result] Dalle Carbonare L, Valenti MT, Del Forno F, Piacentini G, Pietrobelli A. Vitamin D Daily versus Monthly Administration: Bone Turnover and Adipose Tissue Influences. Nutrients. 2018 Dec 6;10(12):1934. doi: 10.3390/nu10121934. PMID 30563215
- [Result] Dalle Carbonare L, Valenti MT, Del Forno F, Caneva E, Pietrobelli A. Vitamin D: Daily vs. Monthly Use in Children and Elderly-What Is Going On? Nutrients. 2017 Jun 24;9(7):652. doi: 10.3390/nu9070652. PMID 28672793
- [Result] Pecoraro L, Nisi F, Serafin A, Antoniazzi F, Dalle Carbonare L, Piacentini G, Pietrobelli A. Vitamin D Supplementation in the Assessment of Cardiovascular Risk Factors in Overweight and Obese Children. Med Sci (Basel). 2022 Sep 5;10(3):49. doi: 10.3390/medsci10030049. PMID 36135834
- [Result] Valenti MT, Pietrobelli A, Romanelli MG, Franzolin E, Malerba G, Zipeto D, Mottes M, Dalle Carbonare L. Molecular and Lifestyle Factors Modulating Obesity Disease. Biomedicines. 2020 Mar 1;8(3):46. doi: 10.3390/biomedicines8030046. PMID 32121611